CLINICAL TRIAL: NCT02336854
Title: Tacrobell tab_Phase1_PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 111HPS14027
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2015-01

CONDITIONS: Immunosuppressant(Organ Transplantation, RA)
Keywords: pharmacokinetics

ARMS (2):
- Tacrobell tab. 2mg (Experimental): 2mg/tablet, PO, 1 tablet once daily for Period I & II D1(crossover)
  Interventions: Drug: Tacrobell tab. 2mg
- Prograf cap. 2mg (Active Comparator): 1mg/capsule, PO, 2 capsule once daily for Period I & II D1(crossover)
  Interventions: Drug: Prograf cap. 2mg

INTERVENTIONS:
Drug: Tacrobell tab. 2mg
  Arms: Tacrobell tab. 2mg
Drug: Prograf cap. 2mg
  Arms: Prograf cap. 2mg

SUMMARY:
A randomized, open-label, two-way crossover study to assess the tolerability and pharmacokinetics of Tacrobell® Tab. and Prograf® Cap. after a single oral dose in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the requirements of the study and voluntarily consent to participate in the study.
2. Healthy male volunteer in the age between 20 and 45 years old.
3. Body weight ≥ 55 kg and 30.0kg/m2 ≥ BMI ≥ 18.0kg/m2

Exclusion Criteria:

1. presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, hematological, gastrointestinal, neurological, psychiatric or other diseases
2. any chronic disease which might interfere with resorption, distribution, metabolism or excretion of the drug, or major surgery of the gastrointestinal tract except for appendectomy
3. any history of drug hypersensitivity (especially to the active and inactive ingredients of the tacrolimus preparation)
4. administration of cyclosporine or Bosentan
5. administration of potassium sparing diuretic
6. Subjects with galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
7. SBP > 150 mmHg or< 90 mmHg
8. DBP > 100 mmHg or < 50 mmHg
9. positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies, RPR
10. AST or ALT > 1.5*ULN, e-GFR < 80 mL/min
11. history of drug abuse or positive drug screening test
12. intake or administration of any ethical or herbal medication medication within 2 weeks, intake or administration of any OTC or vitamin preparations
13. medication with metabolizing enzyme inducers or inhibitors such as barbitals within 1 month before first dosing
14. administration of another study medications within 3 months before first dosing
15. blood donation in 2 months, component blood donation within 1 month or blood transfusion before first dosing
16. Alcohol > 21 units/week or cannot stop drinking during the study
17. Cigarette > 10 cigarettes/day or cannot stop smoking during hospitalization
18. consumption of beverages or food containing caffeine(e.g.coffee, tea) during hospitalization
19. consumption of grapefruit or food containing grapefruit during hospitalization
20. Not eligible to participate for the study at the discretion of investigator.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2015-02-02 (Actual); Study Completion 2015-03-19 (Actual)

PRIMARY OUTCOMES:
AUClast | up to 96 hous postdose
Cmax | up to 96 hous postdose

SECONDARY OUTCOMES:
AUCinf | up to 96 hous postdose
Tmax | up to 96 hous postdose
t1/2 | up to 96 hous postdose
CL/F | up to 96 hous postdose